CLINICAL TRIAL: NCT06717828
Title: The Effects of Tai Chi on Metabolic Dysfunction-associated Fatty Liver Disease in Middle-Aged and Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Xiling lLIN, Associate chief physician, Fujian Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 202410081053000483865
Record Dates: First submitted 2024-12-01; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: MAFLD; Tai Chi; Intrahepatic Fat Content
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Aquatic Therapy

STUDY DESIGN:
Intervention Model Description: The study design utilizes an open, randomized, parallel, controlled approach. A total of 250 middle-aged and elderly subjects with metabolic associated fatty liver disease are recruited. Participants are randomly assigned in a 2:2:1 ratio to the Tai Chi group, conventional exercise group, and control group, with the entire intervention period lasting for 6 months.
Who Masked: Outcomes Assessor
Masking Description: All subjects will undergo all the prescribed baseline assessments before being randomized into groups. The personnel conducting the clinical endpoint assessments will be blinded; they will not be aware of the trial group assignments of the subjects during the measurement of clinical endpoints.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tai Chi Exercise (Experimental): Tai Chi Exercise program, five times a week .
  Interventions: Behavioral: Tai Chi Exercise
- Regular Physical Activity (Experimental): Each exercise session lasts for 60 minutes, five days a week.
  Interventions: Behavioral: Regular Exercise
- Control (Other): Conduct health education on fatty liver once every two months.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Tai Chi Exercise — Tai Chi is a moderate-intensity exercise suitable for middle-aged and elderly individuals. Participants will engage in the practice five times a week (three sessions will be in-person teaching, and two will be online), with each session lasting 60 minutes, continuing until the end of a six-month follow-up. Before the intervention begins, participants will receive a manual or instructional video on Tai Chi to understand its principles, practice techniques, and safety precautions. Each class will start with a warm-up and include a review of Tai Chi principles and movements, breathing techniques, and relaxation methods. Participants will document their Tai Chi practice over 24 weeks by submitting exercise weekly logs, while researchers will monitor their exercise progress weekly via phone using standardized forms to assess frequency, completion status, adverse events, and adherence.
  Arms: Tai Chi Exercise
Behavioral: Regular Exercise — The intervention for middle-aged and elderly individuals includes a combination of common activities: 15 minutes of walking, 15 minutes of body coordination activities (including limb movements and balance training), 15 minutes of muscle stretching, and 15 minutes of relaxation. Each exercise session lasts for 60 minutes, conducted five days a week. The heart rate during exercise will be adjusted based on monthly fitness assessments, and the daily activity level will be evaluated through logs and fitness trackers.
  Arms: Regular Physical Activity
Behavioral: Control — All participants will be advised not to change their existing lifestyle habits and will only receive health education related to fatty liver throughout the intervention. The educational methods will include large group sessions, individual education, and telephone follow-ups, conducted every two months. Additionally, dietary and exercise assessments will be carried out during the intervention, with dietary intake recorded using a three-day food diary to track daily calorie consumption.
  Arms: Control

SUMMARY:
Background: Metabolic dysfunction-associated fatty liver disease (MAFLD) is a liver condition primarily driven by metabolic dysfunctions that may progress to hepatitis, cirrhosis, and hepatocellular carcinoma. It is also implicated in the development of other metabolic dysfunction-related diseases. MAFLD has emerged as a growing public health concern in China. Despite its potential benefits, Tai Chi exercise has not been widely adopted for individuals with MAFLD, and there is limited research investigating its therapeutic efficacy. This study aims to evaluate the effects of a structured Tai Chi intervention on middle-aged and elderly individuals with MAFLD.

Methods: The study employs a comprehensive open, randomized, parallel, and controlled design. Eligible participants will be randomly allocated into three groups: Tai Chi, conventional exercise, and control. A total of 250 participants will be enrolled, comprising 100 participants each for the Tai Chi and conventional exercise groups and 50 for the control group. Both the Tai Chi and conventional exercise groups will participate in a structured 6-month exercise program. During the intervention, both groups will also receive regular health education on fatty liver disease. Participants will be encouraged to maintain their usual activities but will be advised against starting new exercise regimens. The control group will receive only health education on fatty liver disease. The primary efficacy endpoint is the change in hepatic triglyceride content measured via validated imaging techniques after 6 months. Secondary endpoints include changes in total body fat, waist circumference, body weight, blood pressure, blood lipids, blood glucose, insulin sensitivity, pancreatic beta-cell function, kidney function, and pulse wave velocity. Outcomes will be assessed at baseline and post-intervention.

Discussion: Tai Chi exercises demonstrate therapeutic potential in reducing intrahepatic fat content, promoting weight loss, and mitigating cardiovascular risk factors. Furthermore, their efficacy appears superior to that of conventional exercise modalities.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 40 and 75 years;
2. Liver fat content measured by mDixon QUANT is ≥5%;
3. Diagnosis of metabolic associated fatty liver disease;
4. Overweight/obesity (BMI ≥ 24 kg/m²);
5. Signed written informed consent.

Exclusion Criteria:

1. Excessive alcohol consumption (definition: in the past 6 months, males have consumed more than 140g of alcohol per week, and females have consumed more than 70g);
2. Fatty liver due to other causes: such as alcoholic fatty liver, acute and chronic viral hepatitis, drug-induced hepatitis, autoimmune hepatitis, etc.;
3. Severe cardiovascular diseases, including myocardial infarction within the past 6 months;
4. Heart failure (NYHA classification: III - IV);
5. Biliary diseases: such as obstructive biliary diseases;
6. Other diseases affecting glucose and lipid metabolism: diabetes, hyperthyroidism, hypothyroidism, Cushing's syndrome, etc.;
7. Poorly controlled blood pressure: SBP ≥ 180 mmHg, DBP ≥ 100 mmHg;
8. Chronic kidney disease or severe renal impairment, defined as serum creatinine of 135 µmol/L (1.5 mg/dL) for males and 110 µmol/L (1.3 mg/dL) for females;
9. Patients unable to communicate normally, such as those with dementia or cognitive impairment;
10. Currently pregnant or planning to become pregnant in the near future;
11. Other conditions preventing participation in follow-up interventions;
12. Other clinical diseases that make participation in exercise unsuitable, such as inability to cooperate with exercise therapy due to severe pain or joint deformities, or the use of medications that may interfere with the assessment of exercise effects (such as corticosteroids, liver protection drugs, etc.), or medications that affect heart rate (such as beta-blockers).

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Determination of Liver Fat Content | Baseline (month 0) to post-training (month 6)
  The liver is scanned using a SIEMENS 3.0T MRI (Magnetom Prisma, Siemens Healthineers, Germany). Participants lie supine, holding breath at end-expiration. A 3D multi-echo water-fat separation gradient echo sequence is used with parameters: TR 9.00 ms, TE1-6 at 1.05-7.38 ms, 4° flip angle, 450×394 mm FOV, 1.4×1.4×3.5 mm voxel size, 64 slices, 13 sec collection time. Images include in-phase, out-of-phase, water, fat, fat fraction, and R2* relaxation. Liver fat content (%) is measured in pseudocolor mode. ROIs are selected in liver's left lobe, central right lobe, and posterior right lobe below the portal vein at two levels, each 4 cm², avoiding bile ducts and vessels. Average fat content from 9 ROIs represents total liver fat content.

SECONDARY OUTCOMES:
Body weight | Baseline (month 0) to post-training (month 6)
  The measurement is conducted in the morning on an empty stomach, with advance notice given to participants.A standardized scale provided by the research center is placed on a flat surface.Participants are required to remove shoes, hats, and outerwear, and to wear only a single layer of clothing, removing any personal items such as wallets and phones.Participants stand calmly on the scale with their feet symmetrically positioned. Their bodies should be upright, arms naturally relaxed at their sides, head straight, and eyes looking forward.Measurements are taken twice, recording the average, ensuring that the discrepancy between the two measurements is less than 1.0 kg, with precision to 0.1 kg. Participants are advised to maintain an upright posture.
Waist circumference | Time Frame: Baseline (month 0) to post-training (month 6)
  Waist circumference is measured in the morning after fasting. Subjects must stand upright with relaxed abdomen, arms down, and feet together. Use a metric tape at the midpoint between the lower ribs and upper iliac crest (about 1 cm above the navel), wrapped snugly but not compressing the skin. Subjects should breathe normally with a relaxed abdomen, and the measurement is taken at the end of exhalation, avoiding abdominal muscle contraction or breath holding. Repeat twice and record the average, ensuring measurements differ by less than 2 cm, accurate to 0.1 cm.
Blood pressure | Baseline (month 0) to post-training (month 6)
  Subjects must avoid heavy exercise, training, eating, drinking (except water), caffeine, extreme temperatures, and blood pressure-altering meds before measuring. Stop smoking 30 min prior. Relax, empty bladder, rest 5 min. Measure BP in a comfortable room, seated naturally with back straight, palms up. Cuff on bare skin, 1-2 cm above inner elbow, not covering joint, tube aligned with middle finger. Cuff center at heart level. After one measurement, loosen cuff, let subject move arm slightly, then rest 1-2 min before next. Take three measurements, 1 min apart, to 1 mmHg precision.
Grip strength of both hands | Baseline (month 0) to post-training (month 6)
  Using a calibrated hand dynamometer (Brand: CAMRY, Model: EH101).Subjects may stand or sit with their upper limbs naturally hanging at their sides. The palm should face the inner side of the body, with the handle of the dynamometer facing outward.Subjects should grip the dynamometer firmly to measure their grip strength, maintaining a stable posture without swinging the dynamometer back and forth during the measurement.Measure three times and record the maximum value. The dynamometer should be reset to zero before each measurement. Values should be recorded with a precision of 0.1 kg. The measurement can be conducted in the order of right hand followed by left hand.
Body fat percentage | Baseline (month 0) to post-training (month 6)
  Using the BIA method, which calculates the proportion of fat and non-fat tissues based on the principle that well-hydrated tissues like muscles and blood vessels conduct electricity well, while fat tissue hardly conducts electricity at all.Measurements should be taken in a fasting state in the morning or more than 2 hours after a meal, with prior notification to the subjects; subjects should avoid vigorous exercise, saunas or baths, excessive alcohol consumption, and the intake of large amounts of water or food (1-2 hours before).Place the body fat analyzer (InBody 770, provided by the research center) on a flat, hard surface. The subject should stand barefoot on the foot electrodes of the body fat analyzer with dry skin, straighten the back and knees, raise the arms horizontally, extend the elbows, and position the arms at a 90° angle from the body with the palms pressed against the electrodes.Precision is to 0.1%.
Total body fat | Baseline (month 0) to post-training (month 6)
  To measure total body fat, a DEXA densitometer scans subcutaneous fat and body composition. Subjects wear minimal clothing, remove metals, and lie centered on the scanning bed, aligned with the midline. For wider bodies, a half-body scan is possible. The scan includes the head, spine, and one side of the body, with the head 3 cm below the bed's horizontal line. Hands are positioned thumbs up, palms to legs, and arms alongside the body. Nylon straps secure knees and feet. Start the scan from the toolbar, monitor the image for full body display, and reposition if needed. Composition results show fat percentage, and detailed reports are printed from the Reports dialog box.
Liver fibrosis scanning to determine liver stiffness | Baseline (month 0) to post-training (month 6)
  The FibroScan PRO-S by Echosens measures liver elasticity to assess hardness. Subjects lie supine with the right arm extended. Operators sit on the right, facing the subject and screen, placing the probe between ribs near the liver's right lobe, avoiding the edge. Use A-mode and M-mode to find a 6 cm deep, vascular-structure-free area, keeping the probe perpendicular to the skin. Press until the pressure indicator is green, then press the probe button for 1/10 sec data acquisition. Check the elastogram quality. For disinfection, end the exam, wipe off gel, and clean the probe tip with an alcohol-free disinfectant. Calibrate the probe every 12 months.
Abdominal visceral fat | Baseline (month 0) to post-training (month 6)
  Abdominal visceral fat measurement is performed using the SIEMENS 3.0T MRI instrument (Magnetom Prisma, Siemens Healthinners, Erlangen, Germany). During the examination, subjects lie in a supine position and hold their breath while a single-layer cross-sectional MRI scan is taken at the L4-L5 level. After the acquisition, Image J software is used to analyze the area of abdominal visceral fat.
Blood specimen | Baseline (month 0) to post-training (month 6)
  Lab tests include OGTT at 0, 30, 120 min, serum insulin at 0, 30, 120 min, HbA1c, lipids, liver and kidney function. Fasting blood is collected early morning by trained nurses. For OGTT (7-9 a.m.), subjects fast 8-10 hours and drink 75g anhydrous glucose in 300ml water (or 82.5g monohydrate) within 5 min. Blood samples are taken pre-test and at 30, 120 min post-glucose. Avoid tea, coffee, smoking, and heavy exercise. Samples are sent to Fujian Provincial Hospital lab for uniform testing, following standards and accredited.

CONTACTS AND LOCATIONS:
Locations (1):
- Fujian Provincial Hospital, Fuzhou, Fujian, China